CLINICAL TRIAL: NCT02919826
Title: Adapting and Evaluating Dialectical Behaviour Group Therapy for Adults With Dual Diagnosis (Intellectual Disabilities With Psychiatric Disorder)
Brief Title: Dialectical Behaviour Group Therapy for Adults With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Jessica Jones (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Sponsor-Investigator, Dr. Jessica Jones, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSIY-511-15
Record Dates: First submitted 2016-09-12; First posted 2016-09-29 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DBT Group (Experimental): Adapted Dialectical Behaviour Therapy
  Interventions: Behavioral: Adapted Dialectical Behaviour Therapy
- Control Arm (No Intervention): People in this group will receive treatment as usual

INTERVENTIONS:
Behavioral: Adapted Dialectical Behaviour Therapy — 12 weekly sessions of DBT group therapy
  Arms: DBT Group

SUMMARY:
To determine the feasibility and effectiveness of a RCT of an adapted DBT group delivered to individuals with ID and emotional dysregulation.

DETAILED DESCRIPTION:
1.2 Introduction

This pilot intervention attempts to deliver and evaluate an adapted Dialectical Behavior Therapy (DBT) in group format. It is hypothesized that the strategies taught through this adapted modality will increase adults with dual diagnosis skills in managing difficult situations and their emotional reactions, thereby decreasing risk of crisis and ultimately demands placed on the mental health service system.

1.3 Research Questions:

Four key questions are addressed within this project:

1. Can adults with intellectual disabilities learn and retain knowledge and skills presented in an adapted DBT group program?
2. Do participants report positive increases in self-esteem and greater engagement in social situations following group participation?
3. Are there decreases in signs and symptoms of mental health issues i.e. anxiety and depression and improvements in challenging behavior following completion of the dialectical behavior group therapy program?
4. Does the program provide any benefit to caregivers? (e.g., are the able to de-escalate "crisis" situations quicker? Do caregivers feel it provides them tools to use when the client experiences distress? Does it lessen the caregivers stress?)

2. Methods

2.1 Research Design:

Building upon the DBT adaptation work performed in the United States by Charleton and Dykstra (2011), it is necessary to further refine this intervention to increase its feasibility and viability as a treatment modality for the adult population with dual diagnosis. Using a mixed-methods approach within this current intervention allows exploration of DBT group therapy efficacy for adult with ID and emerging mental health/behavioural issues.

2.2 Recruitment:

Participants and caregivers will be invited to participate through the use of local advertising at partnering agencies and through expression of previous interest to clinicians involved. Information brochures/flyers will be distributed to individuals who have expressed an interest in counseling services and may or may not be receiving services at the time. Once participants have been identified they will have the opportunity to self-select a caregiver who they would like to assist them in the groups. The caregivers will receive a letter of information and consent form requesting their participation. All participants will be screened for eligibility and attainment of consent for involvement will include the use of a multi-modality approach.

Agencies to be recruited: Ongwanada, Providence Care MHS DDCOT, Christian Horizons, Community Living Kingston, Developmental Services Leeds and Grenville (DSLG), Pathways

2.3. Procedure

1. Recruit
2. Screen for Eligibility
3. Obtain Written Consent (to be confirmed at Pre-Assessment)
4. Complete Pre-Assessment and confirm informed Consent

   a. At acceptance into the study, individuals will be assigned alpha-numeric symbols on all data documents to ensure patient confidentiality and ensure individuals are unidentifiable to research team. Individuals will be encouraged to use first names only during group sessions and all identifiers (name tags, sign in sheets) will be destroyed at the end of the treatment trial.
5. Once have n=12 participants, Randomize into Group A Intervention or Control
6. Send info package with date/location of group
7. Group A (Duration: 12 weeks)

   a. Divided into 3 modules (Distress Tolerance; Emotion Regulation; Interpersonal Effectiveness, with Mindfulness integrated into each
8. Post Assessment of Group A Participants (n=6) and n=6 new participants
9. Repeat steps 4 to 8 for Group B and C 12-week intervention and control groups.

2.6 Analysis:

Global and individual change question analyses will be conducted within a mixed method approach using SPSS 22. Measures of pre-post group findings will be evaluated using paired t-tests and ANOVAS, if applicable. Structured interview data will be analyzed using thematic analysis where qualitative themes will be summarized and consolidated into possible areas addressing curriculum content, therapeutic process, skill application and overall group therapy feedback

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild or Moderate Intellectual Disability
* Symptoms of emotional and behavioural difficulties e.g. emotional dysregulation
* Dedicated caregiver to accompany and attend all sessions

Exclusion Criteria:

* Diagnosis of Autism Spectrum Disorder
* Profound or Severe Intellectual Disability
* Acute psychosis interfering with daily functioning

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jones, PhD, Principal Investigator — Queen's University, Kingston
Locations (1):
- Division of Developmental Disabilities, 191 Portsmouth Avenue, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DBT Group | Control Arm
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBT Group | Control Arm | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Difficulties in Emotional Regulation Scale (Gratz & Roemner, 2004)
Description: Psychometric measure of emotional dysregulation: Total items 36 (range 36-180), responses ranging from 1 to 5, where 1 is almost never (0-10%), 2 is sometimes (11- 35%), 3 is about half the time (36-65%), 4 is most of the time (66-90%), and 5 is almost always (91-100%). DERS items were recoded so that higher scores in every case indicated greater difficulties in emotion regulation (i.e., greater emotion dysregulation).
Time Frame: Pre treatment and 12 week post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DBT Group Intervention: Adapted Dialectical Behaviour Therapy
  Adapted Dialectical Behaviour Therapy: 12 weekly sessions of DBT group therapy
Arm/Group | DBT Group Intervention | Control Arm
Number analyzed (Participants) | 10 | 8
score on a scale | 1.4 (18.5) | 0.8 (13.2)

2. Secondary Outcome: Change in Novaco Anger Scale: Part B (Provocation Index)(Novaco, 2003)
Description: Psychometric measure of anger dyscontrol as part of total anger scale: Total items 25 (range 25-100), responses ranging from 1 to 4, where 1 is not at all angry, 2 is a little angry, 3 is fairly angry and 4 is very angry. NAS-PI were recoded so that higher scores in every case indicated greater difficulties in anger control (i.e., greater anger dyscontrol).
Time Frame: Pre treatment and 12 week post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DBT Group Intervention: DBT Group Intervention
- DBT Control Group: DBT Control Group will receive treatment as usual.
Arm/Group | DBT Group Intervention | DBT Control Group
Number analyzed (Participants) | 10 | 8
score on a scale | 6.4 (15.6) | 5.6 (11.7)

3. Secondary Outcome: Change in Reiss Scale of Dual Diagnosis 38Q (IDS, 1987)
Description: Psychometric measure of psychiatric illness in individuals with intellectual disabilities: Total items 26 (range 26-78), responses ranging from 1 to 3, where 1 is no problem, 2 is problem and 3 is always a problem. REISS items were recoded so that higher scores in every case indicated greater problems with mental health issues ( i.e. psychopathology.)
Time Frame: Pre treatment and 12 week post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Group Intervention | Control Arm
Number analyzed (Participants) | 10 | 8
score on a scale | 1.8 (9.3) | 2.9 (5.5)

4. Secondary Outcome: Change in Adapted Emotion Regulation Checklist (Adapted With Permission From Dante Cicchetti by Jessica Jones)
Description: Psychometric adapted measure of emotional regulation for informants. Given to caregivers to report on changes in observed emotional regulation. Total items 24 (range 24 - 96) responses ranging from 1 to 4, where 1 is never, 2 is sometimes, 3 is often and 4 is almost always. ERC items were recoded so that higher scores in every case indicated greater emotional regulation.
Time Frame: Pretreatment and 12 week post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Group Intervention | Control Arm
Number analyzed (Participants) | 10 | 8
score on a scale | 4.0 (9.9) | 0.5 (7.4)

5. Secondary Outcome: Global Impression of Change: Percentage of Participants Reporting Improvement
Description: Adapted measure of clinical treatment change for informant: Participants were asked for perceived degree of change post group with total overall change; responses ranging from no change (identified problem got worse), to somewhat better (better but no noticeable change), to better (better but the change has not made a significant difference), to moderately better (slight improved difference) to much better (definite improvement and made a significant difference).
  GIC items were collapsed either into two groups: no change or change (somewhat better, better, moderately better and much better); responses were analyzed in percentages in either group.
Time Frame: 12 week Post Treatment
Population: Following team review participants included in intervention group also belonged to control group. Institutional review board required treatment be offered to control group at end of study. Post-treatment data was collected for all participants who participated in the intervention using this measure. There was missing data (2) for treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Group Intervention | Control Arm
Number analyzed (Participants) | 16 | 0
Participants | 12 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks covering data at baseline, 12 week intervention or control arm and follow-up
Description: Adverse events (serious and non-serious) were monitored as per study protocol.
Arm/Group | DBT Group | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT02919826/Prot_SAP_000.pdf